CLINICAL TRIAL: NCT02494778
Title: A Multi-Center, Open-Label Study Evaluating the Safety, Tolerability, and Efficacy of Pridopidine in Patients With Huntington's Disease (Open PRIDE-HD)
Brief Title: A Study Evaluating if Pridopidine is Safe, Efficacious, and Tolerable in Patients With Huntington's Disease
Acronym: Open PRIDE-HD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study served its purpose in providing considerable safety data.
Sponsor: Prilenia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV7820-CNS-20016; 2015-000904-24 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease, pridopidine
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pridopidine (Experimental): The mode of administration is oral. Capsules will be swallowed whole with water. One capsule should be taken in the morning and 1 in the afternoon, 7 to 10 hours after the morning dose. Study drug can be taken irrespective of meals.
  Interventions: Drug: Pridopidine

INTERVENTIONS:
Drug: Pridopidine — 45 mg BID
  Other Names: TV7820

SUMMARY:
The purpose of the study is to collect and assess long term data on the safety, tolerability, and efficacy of pridopidine in patients with Huntington's disease (HD).

ELIGIBILITY:
Inclusion Criteria:

* Pride HD completion within the last 6 months, including 2 week follow up period or patients who transitioned from the Open HART study or patients who complete future safety and efficacy clinical trials of pridopidine. In addition, patients who have already completed their defined study period under Open PRIDE HD global or local amendments and have discontinued treatment with pridopidine will be allowed to re enter the Open PRIDE HD study.
* Women of child bearing potential or male participants: Adequate contraception and birth control
* Good general health

  * other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Similar baseline criteria for ECG, vital signs, cardiovascular system, and renal function to PRIDE HD;
* Similar concomitant medication restrictions to PRIDE HD.

  * other criteria apply, please contact the investigator for more information

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals USA
Locations (46):
- United States (11):
  - Teva Investigational Site 12204, Los Angeles, California
  - Teva Investigational Site 12201, Englewood, Colorado
  - Teva Investigational Site 12196, Washington D.C., District of Columbia
  - Teva Investigational Site 12206, Baltimore, Maryland
  - Teva Investigational Site 12200, Manhasset, New York
  - Teva Investigational Site 12203, New York, New York
  - Teva Investigational Site 12198, Rochester, New York
  - Teva Investigational Site 12211, Winston-Salem, North Carolina
  - Teva Investigational Site 12209, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12208, Salt Lake City, Utah
  - Teva Investigational Site 12210, Richmond, Virginia
- Australia (3):
  - Teva Investigational Site 78055, Caulfield South
  - Teva Investigational Site 78058, West Perth
  - Teva Investigational Site 78057, Westmead
- Austria (2):
  - Teva Investigational Site 33021, Innsbruck
  - Teva Investigational Site 33027, Vienna
- Teva Investigational Site 11036, Toronto, Ontario, Canada
- France (6):
  - Teva Investigational Site 35123, Angers
  - Teva Investigational Site 35122, Créteil
  - Teva Investigational Site 35125, Lille
  - Teva Investigational Site 35124, Marseille
  - Teva Investigational Site 35121, Salouël
  - Teva Investigational Site 35165, Toulouse
- Germany (4):
  - Teva Investigational Site 32408, Berlin
  - Teva Investigational Site 32410, Bochum
  - Teva Investigational Site 32409, Münster
  - Teva Investigational Site 32407, Ulm
- Italy (4):
  - Teva Investigational Site 30083, Florence
  - Teva Investigational Site 30080, Milan
  - Teva Investigational Site 30082, Napoli
  - Teva Investigational Site 30081, San Giovanni Rotondo
- Teva Investigational Site 38059, Leiden, Netherlands
- Poland (4):
  - Teva Investigational Site 53150, Gdansk
  - Teva Investigational Site 53149, Krakow
  - Teva Investigational Site 53148, Poznan
  - Teva Investigational Site 53151, Warsaw
- Russia (3):
  - Teva Investigational Site 50215, Kazan'
  - Teva Investigational Site 50213, Moscow
  - Teva Investigational Site 50214, Nyznij Novgorod
- United Kingdom (7):
  - Teva Investigational Site 34058, Birmingham
  - Teva Investigational Site 34054, Cambridge
  - Teva Investigational Site 34059, Cardiff
  - Teva Investigational Site 34055, Manchester
  - Teva Investigational Site 34061, Newcastle upon Tyne
  - Teva Investigational Site 34056, Oxford
  - Teva Investigational Site 34057, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen S, Waks Z, Elm JJ, Gordon MF, Grachev ID, Navon-Perry L, Fine S, Grossman I, Papapetropoulos S, Savola JM. Characterizing patient compliance over six months in remote digital trials of Parkinson's and Huntington disease. BMC Med Inform Decis Mak. 2018 Dec 20;18(1):138. doi: 10.1186/s12911-018-0714-7. PMID 30572891

RESULTS

PARTICIPANT FLOW:
Groups:
- Pridopidine 45 mg BID: Pridopidine (45 mg) administered as oral capsules, taken twice daily (bid)
Period: Overall Study
Arm/Group | Pridopidine 45 mg BID
Started | 248
Completed | 27
Not Completed | 221
Not completed — Death | 3
Not completed — Other | 173
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 20
Not completed — Lost to Follow-up | 2
Not completed — Noncompliant with study drug admin. | 1

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Arm/Group | Pridopidine 45 mg BID
Number analyzed (Participants) | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 227
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  Canada | 4
  Austria | 18
  Netherlands | 9
  United States | 34
  Poland | 28
  Italy | 34
  United Kingdom | 28
  France | 18
  Australia | 9
  Germany | 32
  Russia | 34
CYP2D6 metaboliser genotype [Count of Participants; unit: Participants]
  Poor metaboliser | 8
  Extensive metaboliser | 214
  Intermediate metaboliser | 25
  Ultra-rapid metaboliser | 1
Neuroleptic use [Count of Participants; unit: Participants]
  Yes | 94
  No | 154
Number of CAG repeats [Mean (Standard Deviation); unit: CAG repeats] | 44.8 (4.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: From signature of the informed consent form through the end of the study, which was defined as Week 106
Time Frame: 106 weeks
Population: All patients enrolled who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Pridopidine 45 mg BID
Number analyzed (Participants) | 248
Participants | 193

2. Secondary Outcome: Change From Baseline in Quantitative Motor (Q-motor) Measurements, Pro-Sup-Inter-Onset-interval-SD-Hand
Description: Q-motor assessments were based on the application of force transducers and 3-dimensional position sensors. The reported parameter is the Pro-Sup-Inter-Onset-interval-SD-Hand, measured in seconds. Positive change from baseline indicates worsening.
Time Frame: Week 52; end of treatment (EOT) which was planned to occur at Week 104
Population: All patients enrolled who received at least 1 dose of study drug and had at least 1 post-baseline UHDRS-TMS assessment.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Pridopidine 45 mg BID
Number analyzed (Participants) | 146
second
  Change from baseline to Week 52 | 0.0 (0.05)
  Change from baseline to EOT | -0.1 (0.01)

3. Secondary Outcome: Change From Baseline in Quantitative Motor (Q-motor) Measurements, Pro-Sup-Peak-Force-CV-Hand
Description: Q-motor assessments were based on the application of force transducers and 3-dimensional position sensors. The reported parameter is the Pro-Sup-Peak-Force-CV-Hand, measured in %. Positive change from baseline indicates worsening.
Time Frame: Week 52; end of treatment (EOT) which was planned to occur at Week 104
Population: All patients enrolled who received at least 1 dose of study drug and had at least 1 post-baseline UHDRS-TMS assessment.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pridopidine 45 mg BID
Number analyzed (Participants) | 146
percentage
  Change from baseline to Week 52 | -2.9 (9.31)
  Change from baseline to EOT | -5.9 (8.05)

ADVERSE EVENTS:
Time Frame: From signature of the informed consent form through the end of the study, which was defined as Week 106
Arm/Group | Pridopidine 45 mg BID
All-Cause Mortality (participants affected / at risk) | 3/248
Serious Adverse Events (participants affected / at risk) | 31/248
Other Adverse Events (participants affected / at risk) | 191/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine 45 mg BID (N=248)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to varios agents (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Huntington's disease (Congenital, familial and genetic disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Chorea (Nervous system disorders) | 3 (3)
Dystonia (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Peripheral nerve palsy (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine 45 mg BID (N=248)
Fall (Injury, poisoning and procedural complications) | 74 (163)
Contusion (Injury, poisoning and procedural complications) | 13 (20)
Weight decreased (Investigations) | 13 (13)
Chorea (Nervous system disorders) | 23 (30)
Headache (Nervous system disorders) | 14 (19)
Insomnia (Psychiatric disorders) | 20 (27)
Anxiety (Psychiatric disorders) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Nasopharyngitis (Infections and infestations) | 29 (36)

LIMITATIONS AND CAVEATS:
This was an open-label extension of study TV7820-CNS-20002. It was terminated on 10 Nov 2017, as it was considered by the sponsor to have served its purpose in providing long-term safety data. Study termination was not based on safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data and results are owned by the sponsor. Results can be used by the institution for internal noncommercial research, education and patient care, and as required under applicable laws and regulations. Other uses require prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02494778/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02494778/SAP_001.pdf